CLINICAL TRIAL: NCT04594122
Title: Safe Food, Fair Food For Cambodia
Brief Title: Good Hygiene Practice Interventions for Safer Pork at Traditional Markets in Cambodia
Acronym: SFFF Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The International Livestock Research Institute (ILRI) (Other)
Collaborators: National Animal Health and Production Research Institute, Cambodia (Unknown); Livestock Development for Community Livelihood Organization, Cambodia (Unknown); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SFFF-RCT2020
Record Dates: First submitted 2020-09-04; First posted 2020-10-20 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2020-10

CONDITIONS: Food Borne Diseases; Food Safety
Keywords: Hygiene Practice; Bacterial Contamination; Traditional Market; Pork Shop; Cambodia
MeSH Terms: conditions — Foodborne Diseases

STUDY DESIGN:
Intervention Model Description: Two groups of pork retailers will be recruited: control group and intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention in this group
- Intervention (Experimental): Hygiene package, training, branding, and certification
  Interventions: Behavioral: Improve hygiene practice of pork sellers

INTERVENTIONS:
Behavioral: Improve hygiene practice of pork sellers — includes 5 keys actions (Handbook) and provision of equipment incentive and training on good hygiene practices, branding, and certification
  Arms: Intervention

SUMMARY:
Safe Food Fair Food for Cambodia (SFFF) is a Feed the Future Innovation Lab project funded by USAID. This 3-year project aims to improve food safety of animal source food (ASF) in Cambodia. SFFF was awarded to the International Livestock Research Institute (ILRI), National Animal Health and Production Research Institute (NAHPRI) and Livestock Development for Community Livelihood Organization (LDC) and in collaboration with Cambodian Ministry of Health CDC and NIPH. Based on the findings and consultations with food safety stakeholders in Cambodia, we have developed a set of interventions to improve hygienic practice and pork safety at the traditional markets in Cambodia. Those interventions will be introduced and tested at retail in six selected provinces using Randomized Controlled Trials (RCT). To ensure compliance of targeted actors (e.g. retailers), participatory methods (e.g. FGD) were used to validate intervention packages. There are two steps of intervention which contain of part 1) Retailer formative research for SFFF Cambodia and 2) Interventions for Good Hygiene Practices for Safer Pork at Traditional Markets.

Part 1. Retailer formative research for SFFF Cambodia: We will implement an intervention package to this trial group and collect biological sampling to determine the hygienic status before and after the intervention. The intervention packages will be developed for SFFF Cambodia in consultation with partners and based on findings of SFFF Cambodia project.

Part 2. Intervention for Good Hygiene Practices for Safer Pork at Traditional Markets: A randomized controlled trial (RCT) intervention will be conducted in 12 markets in 6 provinces. Those provinces were selected based on the prevalence of Salmonella in a market survey study, namely Kampot, Kampong Cham, Kampong Speu, Takeo, Siem Reap, and Phnom Penh. Another 12 markets, in the same provinces, will be used as a control group. In total 24 traditional wet markets will be included in the sampling, by selecting the 4 largest traditional markets in the six provinces with at least 15 pork shops. At each market, 15 pork shops were selected for sampling. The intervention package includes 5 keys actions (Handbook) and provision of equipment incentive (e.g. inox tray, easy-clean surface material), and training on good hygiene practices.

DETAILED DESCRIPTION:
1. Selection of provinces, markets and retailers

   Six provinces were selected including Phnom Penh, Siem Reap, Takeo, Kampong Cham, Kampot, Kampong Speu with the following selection criteria: i) The number of markets in provinces, ii) Salmonella prevalence (above 50%), iii) Population density and risk, urban - rural, iv) Distance from laboratory, v) Compliance of market board and traders, local animal health workers. Phnom Penh had a reported Salmonella prevalence of less than 50% in the recent market study but was included as an urban center with expected high output of pork sells. In each province, four markets which have at least 15 pork shops will be selected. Among those markets, two markets will be assigned for control and trial groups.

   Group of retailers will be chosen from selected markets for the intervention based on their "similarity" (e.g., environment, shop facilities, sells volume) and their compliance to participate. Intervention package includes providing incentive equipment and training on good hygiene practice. Equipment provision comprise: (i) equip the shops with inox trays and advise them to separate raw pork/processed pork and intestines; (ii) In case the surface of the shop is not made from granite or inox, we will provide them with feasible surface cover material; (iii) Apron to retailers with the project logo/brand; (iv)Shop's banner with our logo; (v) Hand washing soap (antibacterial) and dish detergent; (vi) Disinfectant spray (Anolyte).

   Guide retailers to rearrange their shops to suit their own facility and space. Introduce plastic cutting boards for light cut, check currently used wooden cutting boards at shop to advice to use properly. Introduce frequent washing and disinfection of sale place and shop equipment. Washing with dish detergent and disinfection using spray disinfectant (Electrochemically activated water, pH=7). This shall include:
   * Cutting boards. Washing with dish detergent (soap) and water with scrub, then disinfection using spraying bleach. Leave for five minutes then rinse with water (can also be a spray) and let it air dry. At least prior to open or after closing the shop and once in between.
   * Knives. At least prior to open or after closing the shop and once in between.
   * Cloth. Guide how to use cloth. Each shop should have 2-3 cloth to wipe separate surfaces/tools.
   * Table surface. Require retailers to wash and disinfect throughout at the end of selling day; and apply disinfectant spray at the beginning of the selling day. Only retailers with an easy to clean surface (inox, granite or plastic etc.) shall be selected.
   * Training. Introduce frequent washing of hands, at least once within each selling hour, with clean water and liquid soap, and dry by tissue paper. Proper disposal of tissue paper in closed top bin

   For control group: No intervention or training activities for this group but collection of biological samples and observation checklist to determine hygienic status at their shops over three consecutive days.
2. Intervention description

   1. Procedure to introduce the intervention:

      * Introduce and discuss trial with market authorities and vets (as appropriate)
      * Identify potential retailers, discuss and make plan with them
      * Pre- evaluate current knowledge and practice of selected retailers.
      * Procure suitable (shop size) equipment for "trial" retailers
      * Provide training, instructions and guidelines for selected retailers and introduce equipment
      * Monitoring of hygienic practice, sampling and checking practice of retailer
      * Timelines: "Training and equipment" in the 1st week, follow up, and supervise in week 2-4, sampling will be conducted in the fourth week.
      * Summary report, sharing and discussion with trial retailers to re-evaluate their knowledge.
   2. Procedure for sampling and analysis:

      * At each market, 15 of pork vendors will be selected for sampling.
      * From each vendor, one specimen will be purchased approximately 300 to 400 grams each.
      * All pork samples (n=360) from trial and control groups will be tested for total bacteria count (TBC).
      * In addition, a sub-set of 60 cut pork samples of trial group will be also analyzed for Salmonella Yes/No (qualitative), 30 out of 60 of these samples will be quantified for Salmonella concentration using MPN method.

ELIGIBILITY:
Inclusion Criteria:

* Under selected markets
* Selling pork only
* Daily selling
* Voluntary

Exclusion Criteria:

* Out of the age range 18-65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of samples fulfill Cambodian microbiological standards for pork | 16 weeks
  Total bacterial count in pork samples will be measured from both trial and control groups to assess level of compliance with national standards

SECONDARY OUTCOMES:
Change in knowledge of pork retailers | 16 weeks
  There are 8 questions on the knowledge part. Each correct answer is given 1 score. The minimum and maximum scores of each participant are 0 and 8, respectively. The means of knowledge score will be compared to see the difference between the 2 groups.
Change in practice of pork retailers | 16 weeks
  The practice will be observed using a checklist during the selling time of the sampling day. There are 20 items on the checklist. Each appropriate practice is given 1 score per item. Practice score will be ranged from 0 to 20. The difference between the 2 groups will be compared using means of practice score.

CONTACTS AND LOCATIONS:
Overall Officials: Delia Randolph, PhD, Principal Investigator — The International Livestock Research Institute (ILRI)
Locations (1):
- National Animal Health and Production Research Institute, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No
RCT data can be shared for other researchers but not the IPD.

REFERENCES:
- [Background] Dang-Xuan S, Nguyen-Viet H, Unger F, Pham-Duc P, Grace D, Tran-Thi N, Barot M, Pham-Thi N, Makita K. Quantitative risk assessment of human salmonellosis in the smallholder pig value chains in urban of Vietnam. Int J Public Health. 2017 Feb;62(Suppl 1):93-102. doi: 10.1007/s00038-016-0921-x. Epub 2016 Nov 11. PMID 27837223
- [Background] Darapheak C, Takano T, Kizuki M, Nakamura K, Seino K. Consumption of animal source foods and dietary diversity reduce stunting in children in Cambodia. Int Arch Med. 2013 Jul 17;6:29. doi: 10.1186/1755-7682-6-29. eCollection 2013. PMID 23866682
- [Background] Devleesschauwer B, Haagsma JA, Angulo FJ, Bellinger DC, Cole D, Dopfer D, Fazil A, Fevre EM, Gibb HJ, Hald T, Kirk MD, Lake RJ, Maertens de Noordhout C, Mathers CD, McDonald SA, Pires SM, Speybroeck N, Thomas MK, Torgerson PR, Wu F, Havelaar AH, Praet N. Methodological Framework for World Health Organization Estimates of the Global Burden of Foodborne Disease. PLoS One. 2015 Dec 3;10(12):e0142498. doi: 10.1371/journal.pone.0142498. eCollection 2015. PMID 26633883
- [Background] Dror DK, Allen LH. The importance of milk and other animal-source foods for children in low-income countries. Food Nutr Bull. 2011 Sep;32(3):227-43. doi: 10.1177/156482651103200307. PMID 22073797
- [Background] Gilbert M, Conchedda G, Van Boeckel TP, Cinardi G, Linard C, Nicolas G, Thanapongtharm W, D'Aietti L, Wint W, Newman SH, Robinson TP. Income Disparities and the Global Distribution of Intensively Farmed Chicken and Pigs. PLoS One. 2015 Jul 31;10(7):e0133381. doi: 10.1371/journal.pone.0133381. eCollection 2015. PMID 26230336
- [Background] Grace D. Food Safety in Low and Middle Income Countries. Int J Environ Res Public Health. 2015 Aug 27;12(9):10490-507. doi: 10.3390/ijerph120910490. PMID 26343693
- [Background] Grace D, Omore A, Randolph T, Kang'ethe E, Nasinyama GW, Mohammed HO. Risk assessment for Escherichia coli O157:H7 in marketed unpasteurized milk in selected East African countries. J Food Prot. 2008 Feb;71(2):257-63. doi: 10.4315/0362-028x-71.2.257. PMID 18326173
- [Background] Grace D, Dipeolu M, Olawoye J, Ojo E, Odebode S, Agbaje M, Akindana G, Randolph T. Evaluating a group-based intervention to improve the safety of meat in Bodija market, Ibadan, Nigeria. Trop Anim Health Prod. 2012 Sep;44 Suppl 1:S61-6. doi: 10.1007/s11250-012-0208-z. Epub 2012 Aug 7. PMID 22869336
- [Background] Grace D, Olowoye J, Dipeolu M, Odebode S, Randolph T. The influence of gender and group membership on food safety: the case of meat sellers in Bodija market, Ibadan, Nigeria. Trop Anim Health Prod. 2012 Sep;44 Suppl 1:S53-9. doi: 10.1007/s11250-012-0207-0. Epub 2012 Aug 8. PMID 22872520
- [Background] Hoang VM, Tran TA, Ha AD, Nguyen VH. Cost of Hospitalization for Foodborne Diarrhea: A Case Study from Vietnam. J Korean Med Sci. 2015 Nov;30 Suppl 2(Suppl 2):S178-82. doi: 10.3346/jkms.2015.30.S2.S178. Epub 2015 Nov 6. PMID 26617452
- [Background] Kouame-Sina SM, Makita K, Costard S, Grace D, Dadie A, Dje M, Bonfoh B. Hazard identification and exposure assessment for bacterial risk assessment of informally marketed milk in Abidjan, Cote d'Ivoire. Food Nutr Bull. 2012 Dec;33(4):223-34. doi: 10.1177/156482651203300402. PMID 23424888
- [Background] Kruy SL, Soares JL, Ping S, Sainte-Marie FF. [Microbiological quality of " ice, ice cream. sorbet" sold on the streets of Phnom Penh; April 1996-April 1997]. Bull Soc Pathol Exot. 2001 Dec;94(5):411-4. French. PMID 11889944
- [Background] Lay KS, Vuthy Y, Song P, Phol K, Sarthou JL. Prevalence, numbers and antimicrobial susceptibilities of Salmonella serovars and Campylobacter spp. in retail poultry in Phnom Penh, Cambodia. J Vet Med Sci. 2011 Mar;73(3):325-9. doi: 10.1292/jvms.10-0373. Epub 2010 Nov 2. PMID 21060246
- [Background] Makita K, Fevre EM, Waiswa C, Eisler MC, Welburn SC. How human brucellosis incidence in urban Kampala can be reduced most efficiently? A stochastic risk assessment of informally-marketed milk. PLoS One. 2010 Dec 1;5(12):e14188. doi: 10.1371/journal.pone.0014188. PMID 21152072
- [Background] Meng CY, Smith BL, Bodhidatta L, Richard SA, Vansith K, Thy B, Srijan A, Serichantalergs O, Mason CJ. Etiology of diarrhea in young children and patterns of antibiotic resistance in Cambodia. Pediatr Infect Dis J. 2011 Apr;30(4):331-5. doi: 10.1097/INF.0b013e3181fb6f82. PMID 21412204
- [Background] Nguyen-Viet H, Tuyet-Hanh TT, Unger F, Dang-Xuan S, Grace D. Food safety in Vietnam: where we are at and what we can learn from international experiences. Infect Dis Poverty. 2017 Feb 16;6(1):39. doi: 10.1186/s40249-017-0249-7. PMID 28209208
- [Background] Osbjer K, Boqvist S, Sokerya S, Chheng K, San S, Davun H, Rautelin H, Magnusson U. Risk factors associated with Campylobacter detected by PCR in humans and animals in rural Cambodia. Epidemiol Infect. 2016 Oct;144(14):2979-2988. doi: 10.1017/S095026881600114X. Epub 2016 Jun 23. PMID 27334412
- [Background] Otte MJ, Gumm ID. Intra-cluster correlation coefficients of 20 infections calculated from the results of cluster-sample surveys. Prev Vet Med. 1997 Jul;31(1-2):147-50. doi: 10.1016/s0167-5877(96)01108-7. No abstract available. PMID 9234433
- [Background] Robinson TP, Wint GR, Conchedda G, Van Boeckel TP, Ercoli V, Palamara E, Cinardi G, D'Aietti L, Hay SI, Gilbert M. Mapping the global distribution of livestock. PLoS One. 2014 May 29;9(5):e96084. doi: 10.1371/journal.pone.0096084. eCollection 2014. PMID 24875496
- [Background] Ross T, Sumner J. A simple, spreadsheet-based, food safety risk assessment tool. Int J Food Microbiol. 2002 Jul 25;77(1-2):39-53. doi: 10.1016/s0168-1605(02)00061-2. PMID 12076037
- [Background] Slovic P. Perception of risk. Science. 1987 Apr 17;236(4799):280-5. doi: 10.1126/science.3563507.
- See also: Lindahl J, Kakkar M, Mehta P, Deka R and Grace D. 2014." Risks with Urban and Peri-urban Milk Production in India." Presentation at the EcoHealth 2014 conference, Montreal, Canada, August 11-15. — https://cgspace.cgiar.org/handle/10568/42190
- See also: Lapar, M., L, R. Deka, J. Lindahl, and D. Grace. 2014b. "Quality and Safety Improvements in Informal Milk Markets and Implications for Food Safety Policy." — https://cgspace.cgiar.org/handle/10568/65164